CLINICAL TRIAL: NCT04947644
Title: Comparative Study of Ultrasound-guided Continuous Erector Spinae Plane Block Versus Thoracic Epidural Analgesia in Open Nephrectomy for Renal Malignancy: A Randomized Controlled Study.
Brief Title: Ultrasound-guided Continuous Erector Spinae Plane Block Versus Thoracic Epidural Analgesia in Open Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-301-015
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Erector Spinae Plane Block; Thoracic Epidural Analgesia; Nephrectomy
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural analgesia group (Active Comparator): After negative response, 10 ml of 0.25% bupivacaine will be injected as a bolus dose in the epidural catheter in 5ml divided aliquots at 5min intervals, 30 min before the induction of general anesthesia and the patient will be turned to the supine position. Sensory block will be assessed in operated side by loss of pinprick sensation in midclavicular line every 2 min. After 15min, if the sensory block level was still below T5, an additional 5ml bupivacaine was given. Then followed by continuous infusion of bupivacaine 0.125% at a rate of 6 ml/h that will be started before skin incision and the dose was increased in 2 ml/h increments up to 10 ml/h for 24 hours. Rate adjustment according to pain score and side effects
  Interventions: Procedure: Thoracic epidural analgesia
- Ultrasound guided continuous erector spinae plane block group (Experimental): After verifying the correct space with hydrodissection by 5mL of saline 0.9%, lifting erector spinae muscle off the bony shadow of the transverse process, a catheter was inserted was inserted 3 cm beyond the needle tip and 20 ml of 0.25% bupivacaine will be injected as a bolus dose in the epidural catheter in 10 ml divided aliquots at 5min intervals, 30 min before the induction of general anesthesia and the patient will be turned to the supine position. Sensory block will be assessed in operated side by loss of pinprick sensation in midclavicular line every 2 min. After 15min, if the sensory block level was still below T5, an additional 5ml bupivacaine was given. Then followed by continuous infusion of bupivacaine 0.125% at a rate of 6 ml/h that will be started before skin incision and the dose was increased in 2 ml/h increments up to 10 ml/h for 24 hours. Rate adjustment according to pain score and side effects
  Interventions: Procedure: Ultrasound guided continuous erector spinae plane block

INTERVENTIONS:
Procedure: Thoracic epidural analgesia — After negative response, 10 ml of 0.25% bupivacaine will be injected as a bolus dose in the epidural catheter in 5ml divided aliquots at 5min intervals, 30 min before the induction of general anesthesia and the patient will be turned to the supine position. Sensory block will be assessed in operated side by loss of pinprick sensation in midclavicular line every 2 min. After 15min, if the sensory block level was still below T5, an additional 5ml bupivacaine was given. Then followed by continuous infusion of bupivacaine 0.125% at a rate of 6 ml/h that will be started before skin incision and the dose was increased in 2 ml/h increments up to 10 ml/h for 24 hours. Rate adjustment according to pain score and side effects
  Arms: Thoracic epidural analgesia group
Procedure: Ultrasound guided continuous erector spinae plane block — After verifying the correct space with hydrodissection by 5mL of saline 0.9%, lifting erector spinae muscle off the bony shadow of the transverse process, a catheter was inserted was inserted 3 cm beyond the needle tip and 20 ml of 0.25% bupivacaine will be injected as a bolus dose in the epidural catheter in 10 ml divided aliquots at 5min intervals, 30 min before the induction of general anesthesia and the patient will be turned to the supine position. Sensory block will be assessed in operated side by loss of pinprick sensation in midclavicular line every 2 min. After 15min, if the sensory block level was still below T5, an additional 5ml bupivacaine was given. Then followed by continuous infusion of bupivacaine 0.125% at a rate of 6 ml/h that will be started before skin incision and the dose was increased in 2 ml/h increments up to 10 ml/h for 24 hours. Rate adjustment according to pain score and side effects
  Arms: Ultrasound guided continuous erector spinae plane block group

SUMMARY:
There are different case studies about the use of erector spinae block (ESPB ) in nephrectomy, but there are no enough randomized controlled studies about it until now so it will be one of the earliest studies that investigate the effect of ESPB to relief acute postoperative pain in patients undergoing open nephrectomy.

Although ESPB and thoracic epidural analgesia blocks successfully reduced postoperative opioid consumption in previous studies, no study has ever compared their efficacy in postoperative analgesia of adult patients undergoing open nephrectomy under general anesthesia thus in this randomized comparative study we are aiming to fill this gap in the literature.

The aim of this study is to compare the analgesic effect of ultrasound-guided continuous erector spinae plane block versus thoracic epidural analgesia in open nephrectomy for renal cancer patients.

DETAILED DESCRIPTION:
The erector spinae muscle (ESM) is a complex formed by the spinalis, longissimus thoracis, and iliocostalis muscles that run vertically in the back. The ESP block is performed by depositing the local anesthetic (LA) in the fascial plane, deeper than the ESM at the tip of the transverse process of the vertebra. Hence, LA is distributed in the cranio-caudal fascial plane. Additionally, it diffuses anteriorly to the paravertebral and epidural spaces, and laterally to the intercostal space at several levels.

Cadaveric studies was done on ESPB using MRI to evaluate the spread of local anesthetic mixed with gadolinium dye. Showed the spread of injected volume of 30 ml at level of T10 spread between the level of T5 and T12 . Other cadaveric study showed the spread of the dye to thoracic paravertebral space which may explain the visceral analgesic effect of the block.

There are different case studies about the use of erector spinae block (ESPB ) in nephrectomy, but there are no enough randomized controlled studies about it until now so it will be one of the earliest studies that investigate the effect of ESPB to relief acute postoperative pain in patients undergoing open nephrectomy.

Although ESPB and thoracic epidural analgesia blocks successfully reduced postoperative opioid consumption in previous studies, no study has ever compared their efficacy in postoperative analgesia of adult patients undergoing open nephrectomy under general anesthesia thus in this randomized comparative study we are aiming to fill this gap in the literature.

The aim of this study is to compare the analgesic effect of ultrasound-guided continuous erector spinae plane block versus thoracic epidural analgesia in open nephrectomy for renal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class II.
* Patients undergoing open nephrectomy for malignant renal tumors.
* Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.

Exclusion Criteria:

* Patient refusal.
* Local infection at the puncture site.
* Coagulopathies with platelet count below 50,000 or an international normalized ratio >1.6.
* Renal and hepatic insufficiency.
* Unstable cardiovascular disease.
* History of psychiatric and cognitive disorders.
* Patients allergic to medication used.
* Abnormal anatomy of the thoracic region.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-05-14 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption within 24 hours postoperative | First 24 hours postoperatively.
  Rescue analgesia will be provided in the form of intravenous morphine 3 mg with maximum dose of 0.1 mg/kg/dose (max 0.3 mg/kg/day) boluses if the pain score >3. The total amount of morphine given in 24 hours will be recorded for every patient.

SECONDARY OUTCOMES:
Total intra-operative fentanyl consumption. | Intra-operative
  Elevation of heart rate or mean arterial blood pressure ≥ 20% of the baseline will be treated by fentanyl 0.5 μg / kg
The time of first rescue analgesia. | First 24 hours postoperatively.
  Rescue analgesia will be provided in the form of intravenous morphine 3 mg with maximum dose of 0.1 mg/kg/dose (max 0.3 mg/kg/day) boluses if the pain score >3
Pain using Numerical rating scale (NRS) at rest | First 24 hours postoperatively.
  Pain scores using NRS will be recorded in the post anaesthesia care unit , and for the next 24 hours (1, 2, 4, 6, 12 and 24h) postoperatively. Scores (1-3) are considered mild pain, (4-6) moderate pain and (7-10) severe pain.
Pain using Numerical rating scale (NRS) during movement | First 24 hours postoperatively.
  Pain scores using NRS will be recorded in the post anaesthesia care unit , and for the next 24 hours (1, 2, 4, 6, 12 and 24h) postoperatively. Scores (1-3) are considered mild pain, (4-6) moderate pain and (7-10) severe pain.
Changes in Intraoperative heart rate | Intraoperatively
  It will be recorded before injection of the local anesthetics to be defined as a baseline reading and follow up after injection then will be recorded immediately before and after surgical incision and at 30 min intervals intraoperatively.
Changes in Intraoperative mean arterial pressure | Intraoperatively
  It will be recorded before injection of the local anesthetics to be defined as a baseline reading and follow up after injection then will be recorded immediately before and after surgical incision and at 30 min intervals intraoperatively.
Changes in postoperative mean arterial blood pressure | First 24 hours postoperatively.
  It will be recorded immediately postoperative and at 1, 2, 4, 6, 12 and 24 h postoperatively.
Changes in postoperative heart rate | First 24 hours postoperatively.
  It will be recorded immediately postoperative and at 1, 2, 4, 6, 12 and 24 h postoperatively.
Total dose of bupivacaine consumption. | First 24 hours postoperatively.
  In thoracic epidural analgesia group 10 ml of 0.25% bupivacaine will be injected as a bolus dose in the epidural catheter in 5ml divided aliquots at 5min intervals. After 15min, if the sensory block level was still below T5, an additional 5ml bupivacaine was given.
  In erector spinae plane block group 20 ml of 0.25% bupivacaine will be injected as a bolus dose in the epidural catheter in 10 ml divided aliquots at 5min intervals. After 15min, if the sensory block level was still below T5, an additional 5ml bupivacaine was given.
  In both groups:
  Then followed by continuous infusion of bupivacaine 0.125% at a rate of 6 ml/h that will be started before skin incision and the dose was increased in 2 ml/h increments up to 10 ml/h for 24 hours. Rate adjustment according to pain score and side effects
The incidence of various side effects . | Intra-operative and first 24 hours postoperatively.
  such as hemodynamic instability, nausea, vomiting, dural puncture with the needle or the catheter, post dural puncture headache, failed block, unintentional intravascular injection of local anesthetic, local anesthetic toxicity and respiratory depression (respiratory rate <10/minute) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abd elgalil, MD, Principal Investigator — Assistant Lecturer of Anesthesia ,Pain Relief and ICU National Cancer Institute ,Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: one year from after the end of the study.